CLINICAL TRIAL: NCT02700321
Title: A Prospective , Multicenter , Randomized, Controlled, Parallel-group , Open-label Trial Evaluating Benefits of High Flow Nasal Cannula (HFNC) Oxygen for Preoxygenation During Intubation in Non Severely Hypoxemic Patients
Brief Title: Benefits of High Flow Nasal Cannula Oxygen for Preoxygenation During Intubation in Non Severely Hypoxemic Patients
Acronym: PROTRACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0047
Record Dates: First submitted 2016-02-02; First posted 2016-03-07 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Need for Intubation, No Severe Hypoxemia
Keywords: non severely hypoxemic respiratory failure; preoxygenation; crash induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Flow nasal cannula oxygen (HFNC) (Experimental): Patients randomized in "HFNC" group will received a four minutes preoxygenation period with Nasal High Flow Therapy (HFT) Optiflow ®/Airvo® (60 l/mn FIO2 = 1) before orotracheal intubation under laryngoscopy after crash induction.
  Interventions: Device: OPTIFLOW/ AIRVO
- STANDARD high flow Face Mask (HFFM) (Active Comparator): Patients randomized in "Standard face mask" group will received a four minutes preoxygenation period with a standard face mask (15 l/mn) before orotracheal intubation under laryngoscopy after crash induction.
  Interventions: Procedure: STANDARD Face Mask

INTERVENTIONS:
Device: OPTIFLOW/ AIRVO — Patients randomized in "HFNC" group will received a four minutes preoxygenation period with Nasal High Flow Therapy (HFT) Optiflow ®/AIRVO® (60 l/mn FIO2 = 1) before orotracheal intubation under laryngoscopy after crash induction.
  Arms: High Flow nasal cannula oxygen (HFNC)
Procedure: STANDARD Face Mask — Patients randomized in "STANDARD Face Mask" group will received a four minutes preoxygenation period with a standard face mask (15 l/mn) before orotracheal intubation under laryngoscopy after crash induction.
  Arms: STANDARD high flow Face Mask (HFFM)

SUMMARY:
The aim of this study is to determine whether High Flow nasal cannula (HFNC) oxygen is more efficient than the standard High Flow face mask (HFFM) for preoxygenation before orotracheal intubation after crash induction in non severely hypoxemic patients

DETAILED DESCRIPTION:
This study will be designed as followed : patients will be randomized in 2 groups : High Flow nasal cannula "HFNC" or standard High Flow face mask "HFFM".

Patients randomized in "HFNC" group will receive a four minutes preoxygenation period with Nasal High Flow Therapy (60 L/mn , fraction of inspired oxygen (FI02) = 100%) before orotracheal intubation under laryngoscopy after crash induction. After induction and during laryngoscopy, HFNC will be maintained in an attempt to achieve apneic oxygenation.

Patients randomized in "HFFM" group will received a four minutes preoxygenation period with standard face mask (15 L/mn) before orotracheal intubation under laryngoscopy after crash induction. After induction, HFFM will be removed, enabling laryngoscopic vision

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years regardless of the gender
* Requiring orotracheal intubation in intensive care unit
* "No severely hypoxemic respiratory failure" defined as Oxygen Pression (Pa02)/FI02 > 200 mmHg measured in the 4 hours before inclusion

Exclusion Criteria:

* Not the first Intubation during this stay in intensive care unit
* Contraindication to oro-tracheal intubation
* Intubation without anaesthesic rapid sequence induction
* Intubation during cardiac arrest
* Real emergency (as asphyxia) with immediate intubation needed (without time enough for randomization)
* Nasopharyngeal obstacle with contraindication to use Optiflow device
* Patients with a documented Cormack IV exposition before inclusion
* Protected adult
* Pregnancy or breastfeeding
* Lack of consent
* Patient already enrolled in another study that could interfere with the primary objective of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
lowest pulse oxymetry (SpO2) during intubation | From the beginning of the endotracheal intubation procedure (beginning of laryngoscopy, immediately after induction) to completed orotracheal intubation (airway catheterization). Usual duration is inferior to 10 minutes
  This outcome will be assessed from the beginning of the endotracheal intubation procedure (immediately after induction) to the end of orotracheal intubation (airway catheterization) by monitoring the pulse oxymetry

SECONDARY OUTCOMES:
Pulse oximetry | from the beginning of preoxygenation period to the end of intubation procedure. Usual duration is inferior to 15 minutes
number of desaturation events (under 80%) | From the beginning of the endotracheal intubation procedure (beginning of laryngoscopy, immediately after induction) to completed orotracheal intubation (airway catheterization). Usual duration is inferior to 10 minutes)
Reduction in morbi-mortality during the Intensive care Unit stay | from beginning of the preoxygenation period to discharged from intensive care unit (until day 28 for more)
SOFA score | Each day during the 5 first days after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Olivier ZAMBON, MD, Principal Investigator — Nantes University Hospital
Locations (8):
- France (8):
  - Brest hospital, CHU La cavale Blanche, medical intensive care unit, Brest
  - CHD LES OUDOUAIRIES Service de réanimation polyvalente, La Roche-sur-Yon
  - Ch Le Mans, Le Mans
  - Nantes university hospital, hôtel Dieu, Anesthesia intensive care unit, Nantes
  - Nantes University Hospital, Hôtel Dieu, Medical intensive care unit, Nantes
  - Rennes university hospital, Hôpital Pontchaillou, medical intensive care unit, Rennes
  - Nantes University hospital, Hôpital Laennec, pneumology intensive care unit, Saint-Herblain
  - Tours university hospital, hôpital Bretonneau, medical intensive care unit, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guitton C, Ehrmann S, Volteau C, Colin G, Maamar A, Jean-Michel V, Mahe PJ, Landais M, Brule N, Bretonniere C, Zambon O, Vourc'h M. Nasal high-flow preoxygenation for endotracheal intubation in the critically ill patient: a randomized clinical trial. Intensive Care Med. 2019 Apr;45(4):447-458. doi: 10.1007/s00134-019-05529-w. Epub 2019 Jan 21. PMID 30666367